CLINICAL TRIAL: NCT03336489
Title: Evaluation of the Organization of Continuity of Care for Home Hospice Patients by Four Parisian Health Networks
Acronym: DICODOM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: HPD_2016_24
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms; Neurodegenerative Diseases; Terminal Illness
MeSH Terms: conditions — Neoplasms; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Paris, France, home hospice care for terminally ill patients is organized by four "palliative care networks". These networks are responsible for information sharing and coordination of all health care professionals working with the patient. Two different systems are in place to ensure continuity of care outside working hours, in such a setting. In the first system, palliative care specialists from the network are reachable over the phone 24/7 by the patient or its caregivers, whenever needed. In the second system, medical information about the patient, regularly updated by the network's medical team, is available to professionals via a secure website, so that in case the patient requires an urgent medical home visit outside working hours, the visiting physician has access to accurate information.

The study's goal is to compare patient's and caregiver's satisfaction between these two systems of continuity of care.

For that purpose, patients will be taken care of as usual by every palliative care network. In every instance where the patient or caregivers have reached out for medical help through the network's continuity of care system, the patient or caregiver will be called 5 days later by the investigation team to go through a satisfaction questionnaire (Likert scales)

ELIGIBILITY:
Inclusion Criteria:

* Patient has a disease with fatal prognosis and requires palliative care
* Patient lives in Paris, France
* Patient benefits from home hospice care through one of the four official Paris palliative care networks

Exclusion Criteria:

* Pregnant women
* Breastfeeding womed
* Altered cognitive function with a Mini Mental Status below 20
* Patient not able to communicate or not speaking French
* Patient legally not capable of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients newly followed for home hospice care by the four palliative care networks of Paris, France, during the inclusion period (up to the inclusion of 200 patients)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Satisfaction about the response given by the network's continuity of care system | between the first and tenth day after the patient or caregiver activated the network's continuity of care system
  Patient's (or caregiver's) satisfaction about the response given by the network's continuity of care system, after the patient or caregiver activated this system at night time or during week-ends or bank holliday, as measured on a 4-level Likert scale (verbal questionnaire by phone call)

CONTACTS AND LOCATIONS:
Overall Officials: Herve PICARD, MD MSc, Principal Investigator — Clinical Research Department, Rothschild Foundation, Paris (France)
Locations (4):
- France (4):
  - Reseau QUIETUDE, Paris
  - Reseaux ROPE, Paris
  - Reseau ENSEMBLE, Paris
  - Reseaux ParisOuest, Paris